CLINICAL TRIAL: NCT06558669
Title: Effect of Sugarcane Juice on Liver Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pir Mehr Ali Shah Arid Agriculture University (Other)
Responsible Party: Principal Investigator, Naeem Mujahid, Dietitian, Pir Mehr Ali Shah Arid Agriculture University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAURwI
Record Dates: First submitted 2024-08-11; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Liver; Disease, Inflammatory
Keywords: Fresh Sugarcane juice, Liver diseases, Liver health status
MeSH Terms: conditions — Hepatitis; Liver Diseases

STUDY DESIGN:
Intervention Model Description: My study model is Parallel, as I want to check which dose of fresh sugarcane juice has the best effect on liver health status after the consumption of fresh sugarcane juice for 90days, for this, participants has been divided into, one control and three treatments groups
Who Masked: Investigator
Masking Description: The investigator is the individual responsible for overseeing the clinical trial. Masking the investigator means they are unaware of which treatment group participants belong to. This helps prevent bias in data collection, analysis, and interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): There are 100 participants in this arm and will only consume their prescribed medicines.
- Treatment 1 (Experimental): There are 100 participants in this arm who will consume 170mL of fresh sugarcane juice and take their prescribed medicines.
  Interventions: Other: Fresh Sugarcane juice
- Treatment 2 (Experimental): There are 100 participants in this arm who will consume 230mL of fresh sugarcane juice and take their prescribed medicines.
  Interventions: Other: Fresh Sugarcane juice
- Treatment 3 (Experimental): There are 100 participants in this arm who will consume 300mL of fresh sugarcane juice and take their prescribed medicines.
  Interventions: Other: Fresh Sugarcane juice

INTERVENTIONS:
Other: Fresh Sugarcane juice — Fresh sugarcane juice in different doses will be given to liver patients for 90 days
  Arms: Treatment 1; Treatment 2; Treatment 3

SUMMARY:
This study aims to investigate the potential benefits of sugarcane juice on liver health in patients who are suffering from liver-related conditions. We hypothesize that regular consumption of sugarcane juice may improve liver function and alleviate symptoms in patients with liver disease. Patients participating in this study will consume a specified amount of sugarcane juice daily for 90 days, and their liver health will be monitored to assess any improvements. This study could help identify a natural, accessible treatment option to support liver health in patients with liver disease, potentially improving their quality of life.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) is designed to evaluate the impact of sugarcane juice on liver health in patients diagnosed with liver-related conditions, including cirrhosis, hepatitis, and fatty liver disease. The study aims to assess whether sugarcane juice, administered in varying dosages, has a therapeutic effect on liver enzyme levels and overall liver function.

Study Design

This is an interventional study using a randomized controlled trial (RCT) design. Participants will be randomly assigned to one of four groups: three treatment groups and one control group. The treatment groups will receive daily doses of sugarcane juice at 170mL, 230mL, and 300mL, respectively, along with their prescribed medicine, for a duration of three months. The control group will receive no sugarcane juice but will continue their prescribed medication regimen.

Intervention Details

Control Group: Receives no sugarcane juice, only prescribed medication. Group 1: Receives 170mL of sugarcane juice daily along with prescribed medication.

Group 2: Receives 230mL of sugarcane juice daily along with prescribed medication.

Group 3: Receives 300mL of sugarcane juice daily along with prescribed medication.

Duration of the Study

The study will span three months, during which participants' liver health will be monitored at regular intervals.

Outcome Measures

Primary Outcome Measures:

Levels of liver enzymes: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), and Total Bilirubin.

Secondary Outcome Measures:

Changes in liver-related symptoms, including jaundice, abdominal pain, fatigue, and nausea.

Sample Size

The study will enroll a total of 400 participants. The participants will be divided into four groups:

Control Group: 100 participants Group 1: 100 participants Group 2: 100 participants Group 3: 100 participants

Inclusion and Exclusion Criteria

Inclusion Criteria:

Patients diagnosed with liver disease, including but not limited to cirrhosis, hepatitis, or fatty liver disease.

Age group 20-60 years. Symptoms criteria based on liver disease include jaundice, abdominal pain, fatigue, nausea, and elevated liver enzymes (ALT, AST) as per standard diagnostic criteria.

Exclusion Criteria:

Patients younger than 20 years or older than 60 years. Patients with a history of other chronic conditions that may interfere with liver function, such as chronic kidney disease or heart failure.

Patients who have undergone liver transplantation. Patients currently participating in another clinical trial related to liver disease.

Pregnant or breastfeeding women.

Statistical Analysis Plan

The data will be analyzed using SPSS (version 27). A Two-Way ANOVA will be used to compare the effects of different dosages of sugarcane juice on liver enzyme levels across the treatment groups and control group. Post hoc analysis will be conducted using Tukey's Honest Significant Difference (HSD) test to identify specific group differences.

Quality Assurance Measures

Data Validation: Rigorous input checks, automated testing, and manual reviews will be implemented to ensure data accuracy.

Site Monitoring: Real-time monitoring tools will be employed to track site performance and swiftly identify any data issues.

Auditing: Regular audits will be performed to ensure compliance with the study protocol and to maintain the integrity of the data.

Handling Missing Data

Data Imputation: Both simple and advanced methods will be employed to impute missing data, ensuring the robustness of the dataset.

Data Cleansing: Consistency checks and outlier detection methods will be implemented to correct data errors.

User Feedback: Tools will be provided to allow users to report and correct missing or inconsistent data promptly.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with liver disease, Age group 20 to 60years Symptoms criteria based on liver disease include jaundice, abdominal pain, fatigue, nausea, and elevated liver enzymes (ALT, AST) as per standard diagnostic criteria.

Exclusion Criteria:

Patients younger than 20 years or older than 60 years. Pregnant or breastfeeding women Patients who have undergone liver transplantation. Patients with a history of other chronic conditions that may interfere with liver function, such as chronic kidney disease or heart failure.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Liver Health Status | ["1 Month" at study commencement (Phase 1)]
  Liver health status will assessed through liver function tests including, ALT, AST, ALP, and Total Bilirubin in Phase 1.
LIver Health Status | [Termination of Phase 2(intervention period), "3 Month"]
  Liver health status will assessed through liver function tests including, ALT, AST, ALP, and Total Bilirubin in Phase 2 after completion of three month intervention
LIver Health Status | [Termination of Phase 3 (Washout period), "1 Month"]
  Liver health status will assessed through liver function tests including, ALT, AST, ALP, and Total Bilirubin in Phase 3 which is wash-out time

SECONDARY OUTCOMES:
Dietary Pattern Analysis | [Through studyy compeletion, an avaerage of 9 month]
  Dietary patterns will be analyzed using a Food Frequency Questionnaire (FFQ) to evaluate the patients' intake of various food groups. This will include an assessment of the frequency, portion sizes, and overall dietary diversity. The aim is to correlate dietary habits with the study's primary outcomes.
Dietary Pattern Assessment | [Through studyy compeletion, an avaerage of 9 month]
  A Food Frequency Questionnaire (FFQ) will be administered to assess the dietary patterns of the patients. This questionnaire will capture the frequency, portion size, and types of food consumed over the study period. The collected data will be used to analyze the relationship between dietary patterns and the primary outcomes of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Asif Ahmad, Rawalpindi, Punjab Province, Pakistan